CLINICAL TRIAL: NCT03923621
Title: Pilonidal Excision Versus Endoscopic Surgery
Acronym: PEVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Helens & Knowsley Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBN955/V1
Record Dates: First submitted 2019-03-26; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Pilonidal Sinus
Keywords: Endoscopic Pilonidal Sinus Treatment (EPSiT)
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental - EPSiT (Experimental): Endoscopic Pilonidal Sinus Treatment
  Interventions: Procedure: EPSiT
- Control - excision (Active Comparator): Excision treatment
  Interventions: Procedure: Excision

INTERVENTIONS:
Procedure: EPSiT — Specialised fistuloscope to indentify sinus tracts, cautery tracts, remove causative hair, irrigation.
  Other Names: Endoscopic Pilonidal Sinus Treatment
  Arms: Experimental - EPSiT
Procedure: Excision — Surgery to remove all affected tissue, followed by wound closure.
  Arms: Control - excision

SUMMARY:
Compare clinical outcomes of endoscopic pilonidal sinus treatment (EPSiT) with excision treatment with a randomised clinical trial.

DETAILED DESCRIPTION:
Primary outcome: complication rate Secondary outcomes: Quality of life, recurrence rate, length of stay, post operative pain (NRS), return to work time, time to complete wound healing, resource use.

Allocation ratio 2:1

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Pilonidal disease <3 previous treatments
* Previous incision and drainage allowed
* Over 16 years

Exclusion Criteria:

* Co-morbidity >ASA II
* Unable to consent themselves
* Under 16 years
* Vulnerable adults

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-03; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Complication rate | 12 months
  As described by Dindo et al 2004

SECONDARY OUTCOMES:
Quality of life (QoL) | 12 months
  QoL utilising validated tool

CONTACTS AND LOCATIONS:
Locations (1):
- St Helens & Knowsley Hospitals NHS Trust, Prescot, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No